CLINICAL TRIAL: NCT05587400
Title: The Consistency of Cardiac Output Measured by Electrical Cardiometry and Pulmonary Artery Catheter in Cardiac Surgery Patients With Pulmonary Arterial Hypertension or Right Heart Dysfunction
Brief Title: Consistency of Electrical Cardiometry and Pulmonary Artery Catheter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COMEEC
Record Dates: First submitted 2022-09-23; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Pulmonary Arterial Hypertension; Right Ventricular Dysfunction
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Ventricular Dysfunction, Right

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with pulmonary artery hypertension and/or right ventricular dysfunction (Experimental)
  Interventions: Behavioral: passive leg raising; Drug: dobutamine test; Drug: inhaled nitric oxide

INTERVENTIONS:
Behavioral: passive leg raising — transfer a patient from semi-recumbent position to supine position with a 45° leg lifting
Drug: dobutamine test — infusion dobutamine
Drug: inhaled nitric oxide — nitric oxide inhalation

SUMMARY:
Currently, the gold standard method to estimate CO in patients with PAH or RV dysfunction is pulmonary artery catheter (PAC), however, the invasiveness and complexity of PAC has limited its usefulness in many clinical scenarios. By measuring the thoracic electrical bioimpedance, electrical cardiometry (EC) technique has been reported to noninvasively estimate cardiac output (CO) and other parameters related to cardiac contractility and fluid status in various cardiovascular disorders. However, in patients with pulmonary arterial hypertension (PAH) and/or right ventricular (RV) dysfunction, few study has been reported. The aim of this study is to evaluate the agreement between CO measured by PAC as the referenced method and CO measured by EC technique in patients with PAH and/or RV dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* adult cardiac surgery patients
* pulmonary artery hypertension and/or right heart dysfunction
* mechanical ventilation

Exclusion Criteria:

* life threatening arrhythmia
* severe valve regurgitation
* left ventricular ejection fraction less than 30%
* patients with mechanical circulatory support

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
cardiac output by pulmonary artery catheter | 5minutes after the patients was sedated
  measuring cardiac output using pulmonary artery catheter
cardiac output by electrical cardiometry | 5minutes after the patients was sedated
  measuring cardiac output using electrical cardiometry
cardiac output by pulmonary artery catheter | 2 minutes after passive leg raising
  measuring cardiac output using pulmonary artery catheter
cardiac output by electrical cardiometry | 2 minutes after passive leg raising
  measuring cardiac output using electrical cardiometry
cardiac output by pulmonary artery catheter | 15 minutes after termination of passive leg raising
  measuring cardiac output using pulmonary artery catheter
cardiac output by electrical cardiometry | 15 minutes after termination of passive leg raising
  measuring cardiac output using electrical cardiometry
cardiac output by pulmonary artery catheter | 30 minutes after dobutamine infusion
  measuring cardiac output using pulmonary artery catheter
cardiac output by electrical cardiometry | 30 minutes after dobutamine infusion
  measuring cardiac output using electrical cardiometry
cardiac output by pulmonary artery catheter | 30 minutes after termination of dobutamine infusion
  measuring cardiac output using pulmonary artery catheter
cardiac output by electrical cardiometry | 30 minutes after termination of dobutamine infusion
  measuring cardiac output using electrical cardiometry
cardiac output by pulmonary artery catheter | 30 minutes after nitric oxide inhalation
  measuring cardiac output using pulmonary artery catheter
cardiac output by electrical cardiometry | 30 minutes after nitric oxide inhalation
  measuring cardiac output using electrical cardiometry

CONTACTS AND LOCATIONS:
Overall Officials: Guang-wei Hao, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan hospital Fudan University, Shanghai, Shanghai Municipality, China